CLINICAL TRIAL: NCT06308068
Title: A Single Dose, Randomized, Open-label, Two-way Crossover Bioequivalence Study of Diacerein 50 mg Capsule and Reference Product (ARTRODAR®) in Healthy Thai Volunteers Under Fed Conditions
Brief Title: Bioequivalence Study of Diacerein 50 mg Capsule in Healthy Thai Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: International Bio service (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BE24-002
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteer
Keywords: Diacerein 50 mg Capsule
MeSH Terms: interventions — diacerein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Generic diacerein 50 mg capsule (Experimental): Each subject will receive a single dose of generic diacerein 50 mg capsule, EIDAR, as a test formulation (T), or a single dose of diacerein 50 mg capsule, with 240±2 mL of ambient temperature drinking water at 30 minutes after the start of standardized HFHC breakfast. Investigational product will be provided to subject in stainless steel cup and subject will be dosed without touching the tablet. This activity will be followed by a mouth check using a tongue depressor and a flashlight to assess the compliance of dosing. The formulations will be given in a crossover fashion as per the randomization schedule. The dosing processes will be conducted under normal light condition.
  Interventions: Drug: Diacerein 50 mg Capsule
- Diacerein 50 mg capsule, ARTRODAR® (Active Comparator): Each subject will receive a single dose of generic diacerein 50 mg capsule, , ARTRODAR®, as a reference formulation (R), with 240±2 mL of ambient temperature drinking water at 30 minutes after the start of standardized HFHC breakfast. Investigational product will be provided to subject in stainless steel cup and subject will be dosed without touching the tablet. This activity will be followed by a mouth check using a tongue depressor and a flashlight to assess the compliance of dosing. The formulations will be given in a crossover fashion as per the randomization schedule. The dosing processes will be conducted under normal light condition
  Interventions: Drug: Diacerein 50 mg Capsule

INTERVENTIONS:
Drug: Diacerein 50 mg Capsule — Diacerein 50 mg Capsule
  Other Names: Diacerein

SUMMARY:
To determine and compare the rate and extent of absorption of a test formulation with that of a reference innovator formulation when given as equal labeled dose in healthy subjects under fed conditions

DETAILED DESCRIPTION:
This study is conducted to investigate bioequivalence information which is required to ensure therapeutic equivalence of a test product and a reference product as well as to be considered as one aspect of product quality. Bioequivalence is defined as the absence of a significant difference in the rate and extent to which the active ingredient or active moiety in pharmaceutical equivalents or pharmaceutical alternatives becomes available at the site of drug action when administered at the same molar dose under similar conditions in an appropriately designed study.

An open label, randomized, two-treatment, two-period, two-sequence, single oral dose, crossover bioequivalence study in healthy Thai volunteers under fed conditions with at least 7 days washout period between the administrations of investigational products of two consecutive periods.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Thai male or female subjects between the ages of 18 to 55 years
2. Body mass index between 18.5 to 30.0 kg/m2
3. Normal laboratory values, including vital signs and physical examination, for all parameters in clinical laboratory tests at screening Any abnormalities from the normal or reference range will be carefully considered clinically relevant by the physician as individual cases, documented in study files prior to enrolling the subject in this study.
4. Non-pregnant woman (negative pregnancy test) and not currently breast feeding
5. Female subjects abstain from either hormonal methods of contraception (including oral or transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs, postcoital contraceptive methods) or hormone replacement therapy for at least 28 days prior to check-in in Period 1. Injectable contraceptives e.g. Depo-Provera® will be discontinued at least 6 months prior to check-in in Period 1. Subjects agree to use acceptable non-hormonal contraceptive methods such as condom, diaphragm, foams, jellies, or abstinence for at least 14 days prior to check-in in Period 1 until 7 days after the end of study in Period 2. Female subjects of non-childbearing potential must meet at least one of the following criteria prior to check-in in Period 1:

   * Postmenopausal for at least 1 year or
   * Surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) at least 6 months
6. Male subjects who are willing or able to use effective contraceptive e.g. condom or abstinence after check-in in Period 1 until 7 days after the end of study in Period 2.
7. Have voluntarily given written informed consent (signed and dated) by the subject prior to participating in this study

Exclusion Criteria:

1. History of allergic reaction or hypersensitivity to diacerein or rhein or anthraquinone derivatives or to any of the excipients
2. History or evidence of clinically significant renal, hepatic, gastrointestinal, hematological (e.g. anemia), endocrine (e.g. hypo-/hyperthyroid, diabetes), pulmonary or respiratory (e.g. asthma), cardiovascular (e.g. hypo-/hypertension), psychiatric, neurologic (e.g. seizures), allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) or any significant ongoing chronic medical illness
3. Have high risk for coronavirus infection based on risk assessment questionnaire or diagnosed as confirmed case of COVID-19
4. History about administration of COVID-19 vaccine within 30 days prior to check-in in each Period.
5. History or evidence of enterocolic disturbances such as irritable colon
6. History or evidence of inflammatory intestinal disease (e.g. ulcerative colitis, Crohn's disease), intestinal obstruction or pseudo-obstruction, painful abdominal syndromes of undetermined cause
7. History or evidence of severe liver disease
8. History or evidence of galactose intolerance, the Lapp lactase deficiency or glucosegalactose malabsorption
9. History of sensitivity to heparin or heparin-induced thrombocytopenia
10. History of problems with swallowing tablet or capsule
11. Any condition possibly affecting drug absorption e.g. gastrectomy, enterectomy, gastritis or duodenal or gastric ulceration other than appendectomy
12. History of diarrhea or vomiting or dehydration within 24 hours prior to check-in in each period
13. History or evidence of drug addict or investigation with urine sample shows a positive test for drug of abuse (morphine, marijuana or methamphetamine)
14. Investigation with blood sample shows level of potassium less than 3.5 or more than 5.0 mmol/L at screening laboratory test.
15. Have eGFR (CKD-EPI) < 50 mL/min/1.73 m2 based on serum creatinine results, at the screening laboratory test or during enrollment
16. Abnormal liver function, ≥1.5 times of upper normal limit of reference range for ALT, AST or bilirubin levels at screening laboratory test
17. Investigation with blood sample shows positive test for HBsAg
18. History or evidence of habitual use of tobacco or nicotine containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study
19. History or evidence of alcoholism or harmful use of alcohol (less than 2 years) i.e., alcohol consumption of more than 14 standard drinks per week for men and 7 standard drinks per week for women (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 mL of 40% distilled spirits, such as rum, whisky, brandy, etc.)
20. History or evidence of alcohol consumption or alcohol-containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study or alcohol breath test shows positive result In case of alcohol breath test result represents the alcohol concentration range of 1

    - 10 mg% BAC and the physician carefully considers that the value came from other reasons, not from the alcohol drinking behavior of subjects, the test will be repeated two times separately, not more than 10 minutes. The result of the last time should be used for subject's eligibility which must be 0 mg%BAC.
21. History or evidence of habitual consume of tea, coffee, xanthine or caffeine containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study
22. Consume or drink juice of grapefruit or orange or pomelo or its supplement / containing products and cannot abstain for at least 7 days prior to check-in in Period 1 and continued for entire duration of the study
23. Use of prescription or nonprescription drugs (e.g. paracetamol, digoxin, digitoxin, amoxicillin/clavulanic acid, other antibiotics, diuretics, cardiac glycosides, laxative drugs, antacids and chemotherapy), herbal medications or supplements (e.g. St. John's wort), vitamins or mineral (e.g. iron) or dietary supplements within 14 days prior to check-in in Period 1 and continued for entire duration of the study
24. Participated in other clinical trials within 90 days prior to check-in in Period 1 (except for the subjects who drop out or withdrawn from the previous study prior to Period 1 dosing) or still participates in the clinical trial or participates in other clinical trials during enrollment in this study
25. Blood donation or blood loss ≥ 1 unit (1 unit is equal to 350-450 mL of blood) within 90 days prior to check-in in Period 1 or during enrollment
26. Subjects with poor venous access or intolerant to venipuncture
27. Unwilling or unable to comply with schedule visit, treatment plan and other study procedures until end of study
28. Inability to communicate well (i.e. language problem, poor mental development, psychiatric illness or poor cerebral function) that may impair the ability to provide written informed consent or cooperate with clinical team

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2024-08-03 (Estimated); Study Completion 2024-08-18 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax period | Through 36 Hours Post Dose]
  Bioequivalence based on Cmax period
Bioequivalence based on AUC parameters | Through 36 Hours Post Dose]
  Bioequivalence based on AUC parameters

CONTACTS AND LOCATIONS:
Overall Officials: Porranee Puranajoti, Ph. D, Principal Investigator — International Bio service

IPD SHARING:
Plan to Share IPD: No
Confidential